CLINICAL TRIAL: NCT03592186
Title: Adolescents With Substance Use Disorders Transitioning From Residential Treatment to the Community: Improving Outcomes Via a Computer Assisted Parenting Program
Brief Title: Adolescents With Substance Use Disorders Transitioníng From Residential Treatment to the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1802001981; R34DA039289 (NIH)
Record Dates: First submitted 2018-04-25; First posted 2018-07-19 (Actual); Results first posted 2020-12-11 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Substance Use; Adolescent Behavior
Keywords: adolescent; substance use
MeSH Terms: conditions — Substance-Related Disorders; Adolescent Behavior | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parenting Wisely+ (Experimental): Parenting Wisely+ consists of access to the Parenting Wisely computer program (www.parentingwisely.com), paired with engagement strategies: up to four in-person coaching sessions, daily text messages, and access to an online networking forum.
  Interventions: Behavioral: Parenting Wisely+; Behavioral: Treatment as Usual
- Treatment as Usual (Active Comparator): The active comparator is defined as residential treatment services as usual.
  At short-term facility, average length of stay was 6-10 days. At long-term facility, average length of stay was 30-45 days.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Parenting Wisely+ — Parenting Wisely+ experimental intervention
  Other Names: Parenting Wisely; PW
  Arms: Parenting Wisely+
Behavioral: Treatment as Usual — Treatment as Usual

SUMMARY:
Adolescents with substance use disorders (ASUD) in residential treatment have the most serious substance use disorders and the highest rates of psychological, motivational, behavioral, legal, environmental, and vocational problems. ASUD in residential treatment are also at high risk of relapse, with follow-up studies suggesting that 60% of ASUD will relapse within 90 days of discharge. Parenting practices have been established as a key influence on adolescents' initiation and maintenance of substance use, as well as their substance use outcomes and likelihood of relapse. However, therapists who treat ASUD have reported a myriad of systemic barriers to engaging parents in treatment. Findings such as these deem ASUD in residential treatment a high priority population and argue for the value of easily accessible parenting interventions during this critical time. The proposed study evaluates a low cost, low intensity model for delivering parenting skills to parents preparing for their adolescent's discharge from residential substance use (SU) treatment. Specifically, this project involves adapting the delivery of a computerized parenting intervention (Parenting Wisely; PW) that has preliminary evidence of efficacy in improving parenting skills and reducing youth behavior problems. This study adapts the delivery of PW for a new population (parents of ASUD) and new setting (residential treatment), and obtains initial data on its feasibility, acceptability, and effectiveness. As a first step, an open trial with 10 parents was conducted to develop and pilot an adapted version of PW that included moderate engagement strategies: in-person coaching sessions, daily text messages containing reminders of parenting skills and links to video vignettes, and an online parent forum containing two networking boards (Ask an Expert and Connect with Parents). In the current phase, a pilot randomized trial with 60 parents will compare an adapted PW plus treatment as usual (TAU) condition (PW+) versus TAU only in a residential treatment center. Both treatment conditions will be delivered by Bachelor's or Master's-level community clinicians. This small trial will provide some initial evidence regarding the utility of a low-cost, low-intensity intervention and whether a larger, fully powered trial is indicated in the future.

DETAILED DESCRIPTION:
This small pilot trial evaluates a low cost, low intensity model for delivering parenting skills to parents preparing for their adolescent's discharge from residential substance use (SU) treatment. Specifically, this project adapts a computerized parenting intervention (Parenting Wisely; PW) that has preliminary evidence of efficacy in improving parenting skills and reducing youth behavior problems for a new population (parents of adolescents with SU) and new setting (residential treatment).

Participants: A minimum of 60 parent-adolescent dyads will be recruited from residential treatment. To guide design decisions for a larger trial, we made the decision after trial registration to recruit from one short-term residential treatment program and one long-term residential treatment program. Parental inclusion criteria: (1) be parent or legal guardian of an adolescent, aged 12-17 years; (2) had adolescent admitted to residential treatment due to problems related to substance use; (3) will be the primary guardian living with the adolescent immediately post-discharge; (4) willing to receive a parenting intervention; (5) fluent in English or Spanish; and (6) willing to provide written consent. Adolescents qualify if their parents meet these criteria as well as: (1) are fluent in English or Spanish and (2) willing to provide written assent. The only exclusion criteria are conditions that might preclude the adolescent's or parent's participation in a 2-3 hour interview (e.g., mania, psychosis, and cognitive impairment).

Study enrollment and randomization: Parents of all newly admitted adolescents will be screened for substance use and those screening positive, will receive a Consent to Contact (CoC) form. Parents that sign a CoC form will be contacted by research staff and invited in for a consent session.

Parents will provide written informed consent and adolescents will provide written assent in separate private rooms at the residential center. Parents and adolescents may choose to conduct the informed consent process and all study procedures in English or Spanish.

Parents will be given the choice whether to return for the baseline assessment or complete it following informed consent. Randomization will occur within 24 hours after the baseline assessment. Parent-adolescent dyads will be randomized by a blind research staff member to either treatment as usual or PW+ using urn randomization balanced on sex, frequency of substance use, and race/ethnicity. The evaluator will give parents condition assignments in sealed envelopes. If the parent is assigned to PW+, the evaluator will schedule the first coaching session. Coaching sessions were offered via multiple modalities to increase engagement: in-person, phone, or video conference.

Therapist training, fidelity, and competence: Treatment will be delivered by Bachelor's or Master's-level parent coaches, at least one of whom is bilingual in English and Spanish. The study principal investigator (PI) will train the coaches. Coach therapeutic competence will be rated with six items that comprise the "General Therapeutic Skills" section of the Cognitive Therapy Rating Scale (CTRS). A score >24 is the criterion for competence. Study specific adherence checklists have been developed. The coaches will be required to earn a satisfactory consensus CTRS score of >24 and satisfactory adherence ratings (> 80% of elements) on two consecutive role plays to be assigned participants. All sessions will be rated for adherence and competence. A minimum of 25% of tapes will be double rated. The PI will meet weekly with the coaches for supervision focused on how to deliver PW+ with adherence and competence.

Treatment as Usual (TAU): TAU is the standard treatment offered to all patients at the residential center. Adolescents receive about 25 hours of treatment per week with average length of stay 6-10 days at the short-term residential center and 30-45 days at the long-term residential center. Parents are typically offered 2 family therapy sessions. Adolescents receive 4-5 hours of individual and group therapy sessions per day, consisting of psychoeducation and general skills building. Medication management is offered as needed. Prior to discharge, parents also receive standard discharge planning, which consists of either a referral to a new outpatient therapy provider or return to a prior outpatient therapy provider.

Adapted PW program: In addition to TAU , parents in the PW+ will receive: Parenting Wisely online modules, in-person coaching sessions, personalized text messages, and an expert-moderated online parent board.

Parenting Wisely online modules: Parenting Wisely (PW/Ser Padres Con Sabiduría) is a self-administered, interactive, multimedia online program. PW contains video vignettes of ten common family problems (e.g., adolescent substance use, curfews, household chores, monitoring of friends, sibling conflict, improving in school, getting up on time, sharing technology, etc.). For each problem, parents progress through three activities: viewing of a video clip of a family struggling with the problem; selection of one of three possible solutions to the problem; and receipt of feedback about the solution selected. Feedback is presented via a video enactment of the selected solution and an explanation of the solution's pros and cons. Goals of the feedback are to explain why ineffective solutions lead to problems and discuss how effective parenting solutions can prevent and resolve common family issues. Parents receive a parent workbook outlining all 10 vignettes, along with the potential problems and solutions. Parents create a unique login upon enrollment and can complete sessions at their own pace. PW typically takes 3-5 hours to complete.

Individual coaching sessions: Sessions individually tailor PW skills to each parent's presenting concerns, corresponding with four PW vignettes: substance use, limit setting, parental monitoring, and parental communication. The initial session is 60-75 min and consists of three sections: (1) rationale for parenting skills, (2) review of PW substance use module (in session), and (3) practice applying the skill to a current problem. Subsequent sessions follow the same outline and last 45-60 min, with active use of the PW program comprising about half the session. If parents introduce problems/complaints about their adolescent, the coach provides validation and discusses how to apply a pertinent PW skill.

Text-based messaging: Following discharge, parents will receive text messages daily for up to 24 weeks to: (a) reinforce PW skills, (b) motivate continued PW usage, and (c) encourage participation in the online parent message board.

Online parent board: Parents will be given access to a secure, expert-moderated website containing two networking forums (Ask an Expert, Connect with Parents). The website is accessible via a user-friendly smartphone application or "app" (similar to app versions of websites for sites such as Pinterest and Facebook). Parents will be able to submit questions anonymously using the same unique login as for the PW program. Questions posted on the message board will be answered by the research team within 48 hours. Answers to questions posted on the message board will direct parents to a specific PW module(s) most relevant to their parenting question. Participation on the message board will be encouraged for up to 24 weeks post-discharge.

Exit interviews: At each follow-up, parents complete exit interviews containing questions about each aspect of the intervention, including the in-person sessions (e.g., number, content, format), text messages (e.g., content, frequency, format), and online message board (e.g., ease of access, content, format). Parents will also complete the 16-item Consumer Satisfaction Questionnaire (CSQ), which rates their satisfaction with treatment delivery, their adolescent's treatment progress, and their ability to manage their adolescent's problems.

Assessments: Follow-up assessments at 6, 12, and 24 weeks post-discharge will be conducted by an independent evaluator blind to condition. Assessments will be 1.5-2 hours. The primary and secondary outcomes are detailed in the Outcome section. Multiple steps will be taken to prevent attrition. First, multiple sources of contact information will be recorded for parents and adolescents. Follow-up reminders will be made via phone, text, and/or mail. The research team will meet weekly to review no-shows and outreach attempts, and discuss plans to connect with missing participants.

Data analysis plan: All 60 parents will be included in statistical analyses consistent with an intent-to-treat model. Prior to the main analyses, descriptive statistics will be run on key variables to examine distributional properties, identify outliers, and transform variables as needed. The treatment conditions will be compared on baseline demographic and clinical variables using basic two-group independent sample t-tests. Using a p < .05 criterion, significant pre-existing baseline differences between conditions will be controlled in subsequent analyses.

Attrition analyses will compare follow-up completers and non-completers on baseline clinical and demographic variables to determine if they differ systematically. If no systematic differences are found between completers and non-completers, then missing data will be estimated using multiple imputation methods.

Outcomes will be analyzed at 6, 12, and 24 weeks post baseline. Analyses will compare trajectories of use over the post-discharge period, controlling for baseline status as a covariate. For each dependent variable, separate repeated measures Analysis of Covariance will test the influence of condition, controlling for the following covariates: baseline status on the dependent variable, baseline differences between groups, and any mental health or substance use treatment received over the follow-up period. The effect of PW dosage on each dependent variable will be calculated and partial eta squared (η2) will be used to estimate the proportion of variance caused by PW. The primary analytical goal will be to provide measures of association and 95% confidence intervals to reveal the effect size of PW on each dependent variable. The goal of these analyses is to find promising trends to pursue in a larger fully powered trial.

The Primary Aim of the NIH-funded application that funded this study was to establish the feasibility and acceptability of the experimental intervention (Primary Aim 1: To examine the feasibility and acceptability of an adapted PW intervention that includes moderate engagement strategies for parents of adolescents with substance use disorders preparing for discharge from residential). The Secondary Aim of the NIH-funded study was to examine the preliminary effectiveness of the experimental intervention on adolescent substance use, adolescent high-risk behavior, and parenting behavior (Secondary Aims 2-4: To test the effectiveness of the adapted PW intervention + treatment as usual (PW+TAU) versus TAU only on: substance use outcomes, related high-risk behaviors, and parenting skills (the putative mediators of change).) Approximately midway through this study, with the support of the Program Officer, a second residential facility was added. This was to ensure that the study met its pre-specified recruitment targets, and also enabled us to test study procedures at one short-term residential facility and one-long term residential facility, to help inform the design of a future fully powered trial.

ELIGIBILITY:
Inclusion Criteria for Adolescents:

* age 12 years -17 years inclusive
* admitted to residential treatment due to problems related to substance use
* ability to complete study assessments in English or Spanish
* ability to understand and willingness to provide written assent

Exclusion Criteria for Adolescents:

-- Conditions that preclude participation in a 2-3 hour interview (e.g., mania, psychosis, intoxication, cognitive impairment)

Inclusion Criteria for Parents:

* legal guardian of adolescent meeting the adolescent inclusion criteria
* primary custodial guardian of the adolescent after discharge from residential
* access to the internet in the home or workplace to view intervention content, as well as access to a phone that can receive text messages
* ability to complete study sessions and assessments in English or Spanish (and must complete the first baseline assessment prior to teen's discharge from residential)
* ability to understand and willingness to provide written consent

Exclusion Criteria for Parents:

-- Conditions that preclude participation in a 1-2 hour interview (e.g., mania, psychosis, intoxication, cognitive impairment)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara J Becker, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Rosecrance Health Network, Rockford, Illinois
  - Caritas ARTS Program, Cranston, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Individual data will be available upon request to the PI Dr. Sara Becker via email.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Within 6 months of study completion for next 7 years
Access Criteria: Contact the Study PI

REFERENCES:
- [Derived] Becker SJ, Helseth SA, Janssen T, Kelly LM, Escobar KI, Souza T, Wright T, Spirito A. Parent SMART (Substance Misuse in Adolescents in Residential Treatment): Pilot randomized trial of a technology-assisted parenting intervention. J Subst Abuse Treat. 2021 Aug;127:108457. doi: 10.1016/j.jsat.2021.108457. Epub 2021 Apr 30. PMID 34134877

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 74 participants (37 dyads) were recruited from a short-term residential facility and 48 participants (24 dyads) were recruited from a long-term facility.
  The long-term facility was added in Year 3 of the trial to improve recruitment and inform design of a fully powered trial (consistent with recruitment plan outlined in the grant proposal).
Pre-assignment Details: Following informed consent, participants had to complete a baseline assessment and confirm discharge to parental custody (study inclusion criteria) before randomization. 10 participants (5 dyads) that consented were not randomized and not included in the final intent-to-treat sample because of these inclusion criteria.
Units Other Than Participants: Dyads (adolescent + parent)
Groups:
- Parenting Wisely+: Parenting Wisely+ consists of access to the Parenting Wisely computer program (www.parentingwisely.com), paired with engagement strategies: up to four in-person coaching sessions, daily text messages, and access to an online networking forum.
  Parenting Wisely+: Parenting Wisely+ consists of access to the Parenting Wisely computer program, paired with engagement strategies: up to four parent coaching sessions, daily text messages, and access to an online networking forum
  Treatment as Usual: The active comparator is residential treatment as usual
- Treatment as Usual: The active comparator is defined as residential treatment services as usual.
  Treatment as Usual: The active comparator is residential treatment as usual
Period: Overall Study
Arm/Group | Parenting Wisely+ | Treatment as Usual
Started | 60; 30 Dyads (adolescent + parent) | 62; 31 Dyads (adolescent + parent)
6-week Follow-up (At 6-week follow-up, 25 PW+ dyads (25 parents, 24 teens) and 29 TAU dyads (29 parents, 27 teens)) | 49; 25 Dyads (adolescent + parent) | 56; 29 Dyads (adolescent + parent)
12-week Follow-up (At 12-week follow-up, 27 PW+ dyads (25 parents, 22 teens) and 27 TAU dyads (26 parents, 25 teens)) | 47; 27 Dyads (adolescent + parent) | 51; 27 Dyads (adolescent + parent)
Completed (At 24-week (final), 24 PW+ dyads (23 parents, 20 teens) and 27 TAU dyads (25 parents, 26 teens).) | 43; 24 Dyads (adolescent + parent) | 51; 27 Dyads (adolescent + parent)
Not Completed | 17; 6 Dyads (adolescent + parent) | 11; 4 Dyads (adolescent + parent)
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 16 | 11

BASELINE CHARACTERISTICS:
Population: Total number of participants was 122. Analyses were conducted using 61 adolescent-parent dyads, since adolescent and parent data were not independent
Groups:
- Total: Total of all reporting groups
Arm/Group | Parenting Wisely+ | Treatment as Usual | Total
Number analyzed (Participants) | 60 | 62 | 122
Age, Customized [Mean (Standard Deviation); unit: years] — Population: Row population differs from Overall, because age was separately calculated for parents and teens.
  years
    Parent age: number analyzed (Participants) | 30 | 31 | 61
    Parent age | 43.93 (6.52) | 41.23 (6.75) | 42.56 (6.72)
    Teen age: number analyzed (Participants) | 30 | 31 | 61
    Teen age | 15.80 (0.93) | 15.61 (1.12) | 15.7 (1.02)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Teen Female | 15 | 17 | 32
  Teen Male | 13 | 14 | 27
  Teen Other / Prefer not to answer | 2 | 0 | 2
  Parent Female | 26 | 24 | 50
  Parent Male | 4 | 7 | 11
  Parent Other / Prefer not to answer | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Each row separately reports on ethnicity for parents and teens.
  Participants
    Teen Ethnicity: number analyzed (Participants) | 30 | 31 | 61
    Teen Ethnicity: Hispanic or Latino | 10 | 6 | 16
    Teen Ethnicity: Not Hispanic or Latino | 20 | 25 | 45
    Teen Ethnicity: Unknown or Not Reported | 0 | 0 | 0
    Parent Ethnicity: number analyzed (Participants) | 30 | 31 | 61
    Parent Ethnicity: Hispanic or Latino | 8 | 2 | 10
    Parent Ethnicity: Not Hispanic or Latino | 22 | 29 | 51
    Parent Ethnicity: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Data reported for the adolescents in each dyad Population: Each row separately presents racial breakdown for parents and teens. Total number of parents and teens adds up to the total sample
  Participants
    Teen Race: number analyzed (Participants) | 30 | 31 | 61
    Teen Race: American Indian or Alaska Native | 0 | 0 | 0
    Teen Race: Asian | 0 | 1 | 1
    Teen Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Teen Race: Black or African American | 3 | 4 | 7
    Teen Race: White | 21 | 14 | 35
    Teen Race: More than one race | 1 | 8 | 9
    Teen Race: Unknown or Not Reported | 5 | 4 | 9
    Parent Race: number analyzed (Participants) | 30 | 31 | 61
    Parent Race: American Indian or Alaska Native | 0 | 0 | 0
    Parent Race: Asian | 0 | 0 | 0
    Parent Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parent Race: Black or African American | 3 | 5 | 8
    Parent Race: White | 26 | 24 | 50
    Parent Race: More than one race | 0 | 2 | 2
    Parent Race: Unknown or Not Reported | 1 | 0 | 1
Adolescent percent days abstinent over past 90 days (adjusted for days in a controlled environment) [Mean (Standard Deviation); unit: percent] — Population: This analysis was only done with adolescent data. Parents did not report on days of substance use.
  percent
    number analyzed (Participants) | 30 | 31 | 61
    (all) | 58.04 (40.43) | 63.93 (40.49) | 61.03 (40.49)

OUTCOME MEASURES:

1. Primary Outcome: Change in Proportion of Days Used Outside of Controlled Environment
Description: Global Appraisal of Individual Needs - Quick Version (GAIN-Q3) is a well-validated substance use screening tool used to assess adolescent substance use in a range of settings. Substance consumption information is collected using a calendar format with temporal cues (e.g., holidays) to assist in recall of days when alcohol and other drugs were used. Possible number of days range from 0 to 90. Values are adjusted to reflect the proportion of days used outside of controlled environment, with final values ranging from 0 to 1.0; a higher number indicates a higher proportion of days used.
Time Frame: Change from baseline to 24-week post-discharge
Population: This table reports mean values at 12-weeks and 24-weeks with listwise deletion. The pre-specified analytic plan uses mixed models with full maximum likelihood estimation (intent-to-treat) and data from all 30 PW and all 31 TAU adolescents.
Measure: Mean (Standard Deviation); unit: proportion of days used
Arm/Group | Parenting Wisely+ | Treatment as Usual
Number analyzed (Participants) | 30 | 31
proportion of days used
  12 Weeks Post Discharge: number analyzed (Participants) | 22 | 25
  12 Weeks Post Discharge | .27 (.36) | .35 (.41)
  24 Weeks Post Discharge: number analyzed (Participants) | 20 | 26
  24 Weeks Post Discharge | .35 (.36) | .32 (36)
Statistical Analysis 1: Comparison: Parenting Wisely+ vs Treatment as Usual; Mixed models with zero-inflated distributions evaluated whether there was a Time*Condition interaction, using data from the baseline, 12-week, and 24-week assessments. Full maximum likelihood estimation was used. We tested the primary outcome (percent of days of use over the past 90 days, adjusted for time in a controlled environment) for overall number of days of use; Test type: Superiority — In zero-inflated distributions, two outcomes can be specified: 1) probability of being an excess zero (falling outside expected negative binomial distribution), and 2) count value, if not an excess zero. Our focal effect of interest was Time*Condition in the count distribution, i.e. effect of condition over time on predicting the percent of days used greater than zero; p = .12, Mixed Models Analysis; Risk Ratio (RR) = 1.15, 95% CI 2-sided [.97 to 1.36], Standard Error of Mean 2.57

2. Secondary Outcome: Change in Global Appraisal of Individual Needs - Quick Version (GAIN-Q3) Substance-Related Problems Scale
Description: The GAIN-Q3 is a well-validated substance use screening tool used to assess adolescent substance use in a range of settings. The Substance-Related Problems Scale provides a count of substance-related problems experienced over the past 90 days. Possible values range from 0 to 11, with higher scores indicating a greater number of substance-related problems.
Time Frame: Change in substance-related problems from baseline to the 24-week post-discharge assessment
Population: The pre-specified analysis plan uses mixed models with all adolescents randomized to condition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parenting Wisely+ | Treatment as Usual
Number analyzed (Participants) | 30 | 31
score on a scale
  12 Weeks Post Discharge: number analyzed (Participants) | 22 | 25
  12 Weeks Post Discharge | 1.86 (1.89) | 1.36 (1.52)
  24 Weeks Post Discharge: number analyzed (Participants) | 20 | 26
  24 Weeks Post Discharge | 1.40 (1.70) | 1.85 (1.83)
Statistical Analysis 1: Comparison: Parenting Wisely+ vs Treatment as Usual; Mixed models using a linear distribution evaluated whether change in substance-related problems differed by condition. The focal effect was a Time*Condition interaction, using data from the baseline, 12-week, and 24-week assessments. Full maximum likelihood estimation was used; Test type: Superiority; p = .19, Mixed Models Analysis; Risk Ratio (RR) = -.10, 95% CI 2-sided [-.34 to .07], Standard Error of Mean .34

3. Secondary Outcome: Count of Adolescents Testing Negative on Urine Screens
Description: 8 panel urine drug screens testing for marijuana, ecstasy/molly, cocaine, amphetamines, methamphetamines, opiates, oxycodone, and benzodiazepines. Urine screen results will be coded as positive or negative for any substance, and a count of adolescents obtaining a negative urine screen in each condition will be obtained.
Time Frame: 12 weeks
Population: Adolescents who completed a urine screen at 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Parenting Wisely+ | Treatment as Usual
Number analyzed (Participants) | 15 | 20
Participants | 5 | 7
Statistical Analysis 1: Comparison: Parenting Wisely+ vs Treatment as Usual; Comparison of the count of positive urine screens by condition at 12 weeks; Test type: Superiority; p = .92, Chi-squared; Chi-square value = .01

ADVERSE EVENTS:
Time Frame: Approximately 25-30 weeks (baseline assessment done upon admission to residential treatment; follow-ups done over 24 weeks post-discharge. Duration of treatment varied from 6 days to 45 days across the sample)
Description: Used standard National Institutes of Health definition of study-related adverse and serious adverse events.
  Adverse events and serious adverse events were assessed systematically as part of the comprehensive follow-up assessments. Adverse events included instances of juvenile justice involvement (i.e., arrest or incarceration of the adolescent) that were not directly associated with the research, but were temporally associated with the research.
Arm/Group | Parenting Wisely+ | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/62
Other Adverse Events (participants affected / at risk) | 3/60 | 3/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parenting Wisely+ (N=60) | Treatment as Usual (N=62)
Juvenile justice involvement (Investigations) | 3 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
Small pilot trial designed to inform the design of a fully powered trial. The pre-specified analytical plan used mixed models: hence, the outcome values reported here (means, standard deviations) will not align with the primary outcome analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT03592186/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT03592186/ICF_001.pdf